CLINICAL TRIAL: NCT04068090
Title: Taxane Induced Peripheral Neuropathy in Chinese Patients With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: TIPN in China
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, DNA,Peripheral Blood Mononuclear Cells (PBMC)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CIPN: Patients with peripheral neuropathy after treatment with taxanes
  Interventions: Other: Patient Questionnaires; Other: Blood Collection
- Patients without CIPN: Patients treated with taxanes and don't develop will be enrolled to this cohort and matched to a specified subject with neurotoxicity based on age, tumor stage, chemotherapy regimen or total taxane dosage
  Interventions: Other: Patient Questionnaires; Other: Blood Collection

INTERVENTIONS:
Other: Patient Questionnaires — FACT-Ntx, EORTC-CIPN20
Other: Blood Collection — biomarker analysis

SUMMARY:
The purpose of this study is to collect clinical data, blood samples, and self reported symptoms of peripheral neuropathy from Chinese patients with breast cancer after treatment with taxanes. This data will be used to develop predictive markers for neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer
* Females aged 16 and older
* Planning to receive or previous treated with taxanes

Exclusion Criteria:

* Poorly controlled or insulin-dependent diabetes or other condition likely to predispose to neurotoxicity

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chinese breast cancer patients treated with taxanes
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Total score from the FACT-GOG-Ntx questionnaire | Up to 2 years
  Total score from the FACT-GOG-Ntx questionnaire for peripheral neuropathy, ranging from 0-44,higher value represents a worse outcome

SECONDARY OUTCOMES:
Predictive value of genetic variants for the development of neuropathy | In the two weeks before start treatment
  SNPs related to peripheral neuropathy
Total score from the EORTC QLQ - CIPN20 questionnaire | Up to 2 years
  Total score from the EORTC QLQ - CIPN20 questionnaire for peripheral neuropathy, ranging from 20-80,higher value represents a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided